CLINICAL TRIAL: NCT07077369
Title: Phase I Clinical Study of HBx-based mRNA Vaccine (WGc-0201 Injection) Plus Tislelizumab in Hepahepatocellular Carcinoma With High Risk of Recurrence and Metastasis After Radical Therapy
Brief Title: WGc-0201 Plus Tislelizumab in HCC With High Risk of Recurrence and Metastasis After Radical Therapy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jiyan Liu, Deputy Director of the Department of Tumor Biological Therapy, West China Hospital, Sichuan University, West China Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WGc-0201/Tislelizumab -HCC
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- WGc-0201 injection, Dose 1 (Experimental)
  Interventions: Biological: WGc-0201 injection; Drug: Tislelizumab
- WGc-0201 injection, Dose 2 (Experimental)
  Interventions: Biological: WGc-0201 injection; Drug: Tislelizumab
- WGc-0201 injection, Dose 3 (Experimental)
  Interventions: Biological: WGc-0201 injection; Drug: Tislelizumab
- WGc-0201 injection, Dose 4 (Experimental)
  Interventions: Biological: WGc-0201 injection; Drug: Tislelizumab

INTERVENTIONS:
Biological: WGc-0201 injection — WGc-0201 injection
Drug: Tislelizumab — Tislelizumab, 200mg

SUMMARY:
urgical treatment represents a critical approach for HCC patients to achieve long-term survival, primarily including hepatectomy and liver transplantation. With the increasing implementation of HCC screening in China, the proportion of patients eligible for curative-intent surgical resection or ablation has risen annually. However, the 5-year tumor recurrence and metastasis rate post-surgery remains as high as 50%-70%. Postoperative adjuvant therapy has thus become essential to reduce the risk of recurrence and metastasis and improve patient survival. The target population for postoperative adjuvant therapy mainly comprises HCC patients who are suitable for surgical resection but exhibit high-risk factors for recurrence and metastasis. Currently, no internationally standardized adjuvant treatment regimen exists for patients with high postoperative recurrence and metastasis risks. While immunotherapy has demonstrated benefits for advanced HCC, its role in the adjuvant setting is still under exploration.

Hepatitis B virus (HBV) infection is the primary risk factor for HCC, accounting for at least 50% of global HCC cases. In regions with high HBV prevalence-such as East and Southeast Asia, as well as sub-Saharan Africa-the proportion is even higher. While HBV-related HCC can be prevented through vaccination against HBV infection, no specific precision therapy currently exists for patients already diagnosed with HBV-positive HCC. Given that nucleic acid vaccine technology demonstrates value not only in disease prevention but also in immunotherapy-particularly mRNA therapeutic vaccines-this approach holds promise.

mRNA therapeutic vaccines represent a highly promising new modality for tumor treatment. They offer advantages such as excellent safety, long-term expression, and sustained antigen presentation. Additionally, they can mimic the natural infection process of viruses to activate the immune system, eliciting robust immune responses against tumors. Currently, no mRNA therapeutic vaccines targeting HBV-related antigens have been approved for marketing. WGc-0201 Injection is an mRNA therapeutic vaccine encoding HBV-related specific antigens. Its active ingredient consists of modified mRNA encoding HBV-related antigen proteins, formulated into an injectable preparation via lipid nanoparticle (LNP) encapsulation. Preclinical safety evaluations have demonstrated that this vaccine exhibits low toxicity and good tolerability. Building on these preliminary results, this study aims to further evaluate its potential.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed hepatocellular carcinoma (HCC);
* Patients who have undergone curative resection or ablation (limited to radiofrequency ablation [RFA] or microwave ablation [MWA]) within 4-12 weeks prior to enrollment: For those who have undergone curative surgical resection, postoperative pathological examination must confirm negative surgical margins (R0 resection); for those who have undergone ablation, complete radiological response must be demonstrated (complete disappearance of arterial enhancement in all ablated tumor lesions);
* Patients with high-risk factors for recurrence and metastasis following curative resection of HCC;
* Positive for hepatitis B surface antigen (HBsAg);
* No extrahepatic metastasis confirmed by contrast-enhanced CT or MRI either before curative resection or postoperatively.

(Additional inclusion criteria may be supplemented.)

Exclusion Criteria:

* Diagnosed with non-hepatocellular carcinoma such as fibrolamellar carcinoma, sarcomatoid carcinoma, or cholangiocarcinoma mixed with hepatocellular carcinoma;
* Evidence of residual tumor, recurrence, or metastasis;
* Clinically significant ascites;
* Received antitumor treatment after curative resection, excluding a single cycle of TACE (transarterial chemoembolization);
* History of hepatic encephalopathy. (Additional exclusion criteria may be supplemented.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | During one year after initial treatment

SECONDARY OUTCOMES:
Recurrence-Free Survival (RFS) | During two years after initial treatment
Survival rate (2-year and 3-year) | During three years after initial treatment
Safety: Type, frequency, and severity of treatment-related adverse events | During two years after initial treatment